CLINICAL TRIAL: NCT05258825
Title: The Use of Preoperative Monoferric Infusion for Enhanced Recovery After Surgery-driven Elective Abdominal Surgery
Brief Title: Preoperative Monoferric for Abdominal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Pharmacosmos A/S (Industry)
Responsible Party: Principal Investigator, David L., Hepner, MD, MPH, Medical Director, Weiner Center for Preoperative Evaluation, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000761
Record Dates: First submitted 2022-01-13; First posted 2022-02-28 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Anemia; Surgery
MeSH Terms: conditions — Anemia | interventions — ferric derisomaltose

STUDY DESIGN:
Intervention Model Description: This is a single arm study with all study patients receiving intravenous iron infusion.
Masking Description: This is an open label study without masking of participant, care provider, investigator or outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravenous Iron Infusion Arm (Experimental): If the patient is found to have iron deficiency anemia, the patient will receive IV iron preoperatively. Patients that agree to be enrolled in the study will be scheduled for the IV iron dose approximately 3-4 weeks prior to surgery. A single IV dose of 1000 mg of Monoferric will be administered. This will be administered at the Brigham and Women's Hospital infusion center and coordinated with the Hematology team.
  Interventions: Drug: Monoferric

INTERVENTIONS:
Drug: Monoferric — A single intravenous dose of 1000 mg of Monoferric will be administered to a patient 3-4 weeks before anticipated surgery.

SUMMARY:
Although there are multiple formulations of intravenous (IV) iron to choose from, a one-time dose of Monoferric would make it more feasible to integrate it in the perioperative pathway given an often-limited time between preoperative evaluation and surgery date. Furthermore, the one-dose total iron repletion model can offer health economic benefits through reducing red blood cell (RBC) transfusion applying limited resources to establish a perioperative anemia management pathway. Prior studies have described a model that can be used as a baseline which showed cost-savings and outlined each cost component. So far, no US-based approach applying this model has been published.

Hypothesis: Administration of a one-time dose of IV iron to patients with preoperative iron deficiency anemia scheduled to undergo elective abdominal and/or pelvic surgery is feasible. It will result in an increase in preoperative hemoglobin from baseline, and improvement in clinical outcomes.

Aim 1: Determine the change in hemoglobin from baseline after the administration of 1000mg single dose IV iron 3-4 weeks before elective surgery The investigators hypothesize that there will be an increase in hemoglobin levels by 1g/dL by the day of surgery.

Aim 2: Explore the association of IV iron administration on other clinical outcomes including: complications, transfusion of blood products and length of hospital stay.

The investigators hypothesize that there will be a decrease in adverse complications and requirement for transfusion, and shorter hospital stay

Aim 3: Describe the feasibility and process, infrastructure and workflows required to implement an IV iron infusion program

DETAILED DESCRIPTION:
The Food and Drug Administration approved drug Monoferric has a unique structure that allows for a slow, sustained release and bioavailability without free iron toxicity. Efficacy studies demonstrated a faster change in hemoglobin concentration from baseline compared to iron sucrose formulations. The median time to Hb increase of ≥2 g/dL was 28 days. The safety profile was comparable with that of iron sucrose formulations. A previous systematic review reported few hypersensitivity reactions and cardiovascular events among the diverse medical and surgical patient populations.

Although there are multiple formulations of IV iron to choose from, a one-time dose of Monoferric would make it more feasible to integrate it in the perioperative pathway given an often-limited time between preoperative evaluation and surgery date. Furthermore, the one-dose total iron repletion model can offer health economic benefits through reducing RBC transfusion applying limited resources to establish a perioperative anemia management pathway. Prior studies have described a model that can be used as a baseline which showed cost-savings and outlined each cost component. So far, no US-based approach applying this model has been published.

Research design and methods:

The investigators will conduct a single arm clinical trial to measure the change in hemoglobin levels from baseline with the administration of a one-time dose of IV iron to patients with preoperative iron deficiency anemia scheduled to undergo elective major abdominal or pelvic surgery. This prospective study design will allow each participant to function as their own control. The investigators will also describe the infrastructure and workflows required to implement this intervention in the preoperative phase of surgical patient care.

Every patient that is scheduled to undergo a major abdominopelvic surgery will have basic preoperative labs, as a part of standard of care, including a complete blood count during the initial surgical visit. This takes place in the surgeon's outpatient clinic. If the patient's hemoglobin is less than 12 g/dL, reflex iron studies (ferritin and transferrin) will be obtained to diagnose iron deficiency anemia. A serum ferritin level with values below 30 ng per mL or transferrin saturation <20%, consistent with Brigham and Women's Hospital laboratory normal range values, will be used as a cutoff for a positive diagnosis.

Patients that agree to be enrolled in the study will be scheduled for the one-time dose of Monoferric 1000mg intravenous dose approximately 3-4 weeks prior to surgery. This will be administered at the Brigham and Women's Hospital infusion center and coordinated with the Hematology team. The infusion center staff will be administering and monitoring patients receiving the intravenous iron.

Schedule:

1. Week 1: The first visit will be to the surgeon's outpatient clinic (general surgery and gynecology) where the screening process will be initiated. As per standard protocol, hemoglobin labs will be obtained during this initial visit. Anemia related reflex testing will be initiated on these already obtained samples. If the patient meets the laboratory criteria, the nursing assistant will communicate this with the research team.
2. Week 1: If the patient is not available to speak in person, they will be contacted via the phone for consent.
3. Week 1: If the participant is eligible and consented, an appointment will be setup with the Brigham and Women's Hospital infusion center and coordinated by the Brigham Hematology team. This takes place 3-4 weeks before the day of surgery

   1. A single dose infusion of up to 1,000mg Monoferric over a minimum of 20 min until reaching cumulative dosage will be administered. The intravenous iron will be administered at the infusion center by a healthcare professional.
   2. The patient will be monitored for signs and symptoms of hypersensitivity during and after Monoferric administration for at least 30min and until clinically stable following completion of the infusion. Monoferric will only be administered when personnel and therapies are immediately available for the treatment of serious hypersensitivity reactions.
   3. The patient will be provided emergency contact information to report or seek help regarding any concern after they have left the healthcare facility.
4. Week 3 or 4: The patient will arrive the day of surgery to Brigham and Women's Hospital. Hemoglobin labs will be obtained on the day of surgery, in the pre-operative area.

Sample size:

A prior trial of Monoferric in patients with iron deficiency anemia found a mean ± standard deviation change in hemoglobin from baseline to 8 weeks of 2.49 ± 1.30 g/dL, corresponding with a coefficient of variation (standard deviation divided by mean) of approximately 0.5. In the current trial, investigators defined the minimum clinically meaningful change in hemoglobin 3-4 weeks after administration of IV iron in elective surgery patients to be 1 g/dL. Assuming the standard deviation of the change in hemoglobin to be 1.5 g/dL (a conservative three times the coefficient of variation of 0.5 observed in the prior trial), enrollment of 32 patients would provide 95% power to detect a 1 g/dL difference in hemoglobin at a two-sided alpha level of 0.05 using a one-sample t-test.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years old
* Hemoglobin ≤12 g/dL, and ferritin <30ng/mL or transferrin <20%
* Scheduled to undergo elective abdominal/pelvic surgery
* Willingness to participate and sign the informed consent form

Exclusion Criteria:

* Non-iron deficiency anemia
* Hemochromatosis or other iron storage disorders
* Previous serious hypersensitivity reactions to any IV iron compounds
* Treated with intravenous iron within 10 days of IV iron intervention
* Patient has or will be treated with a red blood cell transfusion within 30 days of scheduled surgery
* Received another investigational drug within 30 days of scheduled surgery
* Requiring dialysis or being considered for dialysis
* Already on erythropoietin stimulating agents
* Evidence of decompensated liver cirrhosis or active hepatitis
* Active infection, sepsis
* Alcohol or drug abuse within the past 6 months
* Estimated life expectancy of < 1 year
* Pregnant or nursing women
* Expecting excessive surgical bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Serum hemoglobin concentration | 3-4 weeks after infusion
  change in hemoglobin from baseline after the administration of IV iron

SECONDARY OUTCOMES:
Requirement for perioperative blood transfusion | 1-30 days after surgery
  Explore the association of IV iron administration with perioperative blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Richard D. Urman, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jahn MR, Andreasen HB, Futterer S, Nawroth T, Schunemann V, Kolb U, Hofmeister W, Munoz M, Bock K, Meldal M, Langguth P. A comparative study of the physicochemical properties of iron isomaltoside 1000 (Monofer), a new intravenous iron preparation and its clinical implications. Eur J Pharm Biopharm. 2011 Aug;78(3):480-91. doi: 10.1016/j.ejpb.2011.03.016. Epub 2011 Mar 23. PMID 21439379
- [Result] Auerbach M, Henry D, Derman RJ, Achebe MM, Thomsen LL, Glaspy J. A prospective, multi-center, randomized comparison of iron isomaltoside 1000 versus iron sucrose in patients with iron deficiency anemia; the FERWON-IDA trial. Am J Hematol. 2019 Sep;94(9):1007-1014. doi: 10.1002/ajh.25564. Epub 2019 Jul 13. PMID 31243803
- [Result] Wikstrom B, Bhandari S, Barany P, Kalra PA, Ladefoged S, Wilske J, Thomsen LL. Iron isomaltoside 1000: a new intravenous iron for treating iron deficiency in chronic kidney disease. J Nephrol. 2011 Sep-Oct;24(5):589-96. doi: 10.5301/JN.2011.6248. PMID 21240875
- See also: Company website that manufactures the study drug — https://www.pharmacosmos.com/